CLINICAL TRIAL: NCT05900050
Title: A Phase 2a, Open-label, Randomized, Controlled, Multi-center Proof of Concept Study to Assess the Efficacy, Safety, and Tolerability of VS-01 on Top of Standard of Care, Compared to Standard of Care Alone, in Adult Patients With Acute-on-chronic Liver Failure (ACLF)
Brief Title: Efficacy, Safety and Tolerability of VS-01 in Adult Patients With Acute-on-Chronic Liver Failure and Ascites (UNVEIL-IT)®
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Sponsor Decision
Sponsor: Genfit (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: VS01-IIa-01; 2024-513706-56-00 (EU CTIS Number)
Record Dates: First submitted 2023-06-02; First posted 2023-06-12 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-09

CONDITIONS: Acute-On-Chronic Liver Failure; Ascites
Keywords: Chronic liver diseases; Hepatic Dysfunction; Extrahepatic Organ Dysfunction; Liver Failure; Renal Disease; Hepatic Impairment; Renal Impairment; Hepatic Decompensation; Cirrhosis
MeSH Terms: conditions — Acute-On-Chronic Liver Failure; Ascites; Liver Diseases; Liver Failure; Kidney Diseases; Renal Insufficiency; Fibrosis | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VS-01 on top of SOC (Active Treatment Group) (Experimental): Patients randomized to Active Treatment group will receive VS-01 on top of SOC
  Interventions: Drug: VS-01 on top of SOC
- SOC (Control Group) (Other): Patients randomized to Control group will receive SOC defined as the standard medical management of patients with decompensated cirrhosis and ACLF
  Interventions: Other: SOC (Control Group)

INTERVENTIONS:
Drug: VS-01 on top of SOC — Patients will receive VS-01 intraperitoneally on four consecutive days on top of SOC
  Arms: VS-01 on top of SOC (Active Treatment Group)
Other: SOC (Control Group) — Patients will receive SOC for decompensated cirrhosis and ACLF
  Arms: SOC (Control Group)

SUMMARY:
A Phase 2, multi-center, randomized, controlled, open-label study to evaluate the effects of the intraperitoneal, liposomal formulation VS-01 in patients with an acute episode of hepatic and/or extrahepatic organ dysfunctions and failures in the presence of liver cirrhosis (Acute-on-Chronic Liver Failure, ACLF) and accumulation of fluid in the abdominal cavity (ascites)

ELIGIBILITY:
Inclusion Criteria:

1. Patients with ACLF Grade 1, 2, or 3a according to European Association for the Study of the Liver (EASL)-CLIF criteria;
2. Onset of ACLF not more than 14 days before Baseline (BL);
3. Presence of ascites requiring diagnostic or therapeutic paracentesis;
4. Patients with dry body weight ≥40 and <140 kg;
5. Written informed consent obtained prior to the start of any study-related procedures.

Exclusion Criteria:

1. Presence of any of the following organ failure(s) as per the EASL-CLIF criteria and/or adapted from CLIF-C Organ Failure (CLIF-C OF)/CLIF- Sequential Organ Failure Assessment (CLIF-SOFA) scores:

   1. Respiratory failure necessitating invasive mechanical ventilation;
   2. Coagulation failure (INR > 3.2 or platelet count ≤20 x 109/L);
   3. Severe cardiovascular failure requiring the use of high dose vasopressors;
2. ACLF grade 3b: Presence of four or more organ failures as per EASL CLIF criteria;
3. Presence of spontaneous or secondary bacterial peritonitis;
4. Presence of uncontrolled severe infection(with hemodynamic instability or shock);
5. Poorly controlled seizure disorder;
6. Patients with history of upper gastro-intestinal bleeding over the past 7 days prior to BL, acute bleeding or bleeding upon paracentesis at screening (SCR) or BL;
7. Contraindication for paracentesis;
8. Coagulation disorders such as disseminated intravascular coagulation or hemophilia;
9. Potential or known hypersensitivity to liposomes;
10. Potential or known risk factors for allergic/anaphylactoid like reactions (e.g., mastocytosis/elevated basal tryptase) or multiple hypersensitivities;
11. Patients after organ transplantation receiving immunosuppressive medication;
12. Any severe disease considered to be potentially detrimental at the discretion of the Principal Investigator. This includes but is not limited to hepatocellular carcinoma outside Milan criteria, cholangiocarcinoma, extrahepatic cancer over the past 2 years or people who inject drugs;
13. Need for Renal Replacement Therapy or any extracorporeal liver support device (e.g., MARS®, Prometheus®, plasmapheresis);
14. Alfapump® in place to manage ascites;
15. Pregnancy and lactation;
16. Women of child-bearing potential who are not willing to use adequate contraception;
17. Patients who participate in another clinical trial at the time of SCR or within 4 weeks prior to SCR.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-07-02 (Actual); Primary Completion 2025-10-15 (Actual); Study Completion 2025-10-15 (Actual)

PRIMARY OUTCOMES:
Chronic Liver Failure Consortium (CLIF-C) ACLF score at Day 7 | 7 days

SECONDARY OUTCOMES:
Time to death through Days 28 and 90 | Day 1 through Days 28 and 90
Change in ACLF grade through/at Days 7 and 28 | Day 1 through Day 7 and Day 28, at Days 7 and 28
28-day and 90-day mortality | At Days 28 and 90
Transplant-free survival through/at Days 28 and 90 | Day 1 through Days 28 and 90, at Day 28 and 90
Incidence rate, severity, and relationship to VS-01 of adverse drug reactions and serious adverse drug reactions. | Day 0 to Day 90
  Safety

CONTACTS AND LOCATIONS:
Overall Officials: Pejvack MOTLAGH, M.D, M.Sc, Study Director — Genfit
Locations (26):
- United States (13):
  - University of California Davis Medical Center, Sacramento, California
  - Medstar Georgetown University Hospital, Washington D.C., District of Columbia
  - Tampa General Hospital, Tampa, Florida
  - Piedmont Atlanta Hospital, Atlanta, Georgia
  - Mayo Clinic, Rochester, Minnesota
  - University of Missouri Health Care, Columbia, Missouri
  - Columbia University Medical Center/ New York Presbyterian Hospital, New York, New York
  - Cleveland Clinic, Cleveland, Ohio
  - Medical University of South Carolina, Charleston, South Carolina
  - The Liver Institute at Methodist Dallas, Dallas, Texas
  - Baylor Clinic, Houston, Texas
  - Richmond VA Medical Center, Richmond, Virginia
  - Virginia Commonwealth University, Richmond, Virginia
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- France (4):
  - Centre Hospitalier Régional Universitaire de Tours, Chambray-lès-Tours
  - Hôpital de la Croix Rousse, Lyon
  - Hôpital Universitaire Pitié Salpêtrière, Paris
  - CHU Rennes - Hôpital Pontchaillou, Rennes
- Germany (3):
  - Universitatsklinikum Munster, Münster, North Rhine-Westphalia
  - Charité Universitätsmedizin Berlin, Berlin, State of Berlin
  - Medizinische Hochschule Hannover, Hanover
- Hungary (2):
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Heves Vármegyei Markhot Ferenc Oktatókórház és Rendelőintézet, Eger
- Italy (2):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - Azienda Ospedaliero-Universitaria Policlinico Umberto I, Roma
- Hospital Clínic de Barcelona, Barcelona, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No